CLINICAL TRIAL: NCT05604560
Title: A Neoadjuvant Study of Tislelizumab and SX-682 for Resectable Pancreas Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Lei Zheng (Other)
Collaborators: BeiGene (Industry); Syntrix Biosystems, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Lei Zheng, Executive Director of University of Texas Health Science Center at San Antonio Cancer Center, The University of Texas Health Science Center at San Antonio
Organization: The University of Texas Health Science Center at San Antonio (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTMS 24-0125; STUDY00001055 (Other: University of Texas Health Science Center at San Antonio IRB)
Record Dates: First submitted 2022-10-28; First posted 2022-11-03 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-05

CONDITIONS: Pancreatic Cancer
Keywords: Pancreatic cancer; Adenocarcinoma; Resectable pancreas cancer; Tislelizumab; Anti-PD-1; PD-L1; Antibody; SX-682; CXCR1/2 (chemokine receptor); CXCR1/2 inhibitor; Small molecule; Immunotherapy
MeSH Terms: conditions — Pancreatic Neoplasms; Adenocarcinoma | interventions — tislelizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Arm A - Tislelizumab and SX-682 (Experimental)
  Interventions: Drug: Tislelizumab; Drug: SX-682

INTERVENTIONS:
Drug: Tislelizumab — Patients will receive Tislelizumab (200 mg intravenous) on Day 1 of Cycles 1-6. Cycle 1 will be 14 days long and occur prior to surgery. Cycle 2 will be 14 days long and occur prior to standard of care chemotherapy. Cycles 3-6 will each be 21 days long and will be given after completion of standard of care chemotherapy.
  Other Names: BGB-A317
Drug: SX-682 — Patients will receive SX-682 (200 mg twice daily by mouth) on Days 1-14 of Cycles 1-2 and Days 1-21 of Cycles 3-6. Cycle 1 will be 14 days long and occur prior to surgery. Cycle 2 will be 14 days long and occur prior to standard of care chemotherapy. Cycles 3-6 will each be 21 days long and will be given after completion of standard of care chemotherapy.

SUMMARY:
The purpose of this study is to evaluate the safety and clinical activity of tislelizumab (an anti-PD-1 antibody) in combination with SX-682 (a CXCR1/2 inhibitor) in subjects with newly diagnosed and surgically resectable pancreatic adenocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand and willingness to sign a written informed consent document.
* Age ≥18 years.
* Newly diagnosed have histologically or cytologically proven adenocarcinoma of the pancreas.
* Tumor must be resectable.
* Patient's acceptance to have a tumor biopsy.
* ECOG performance status 0 or 1
* Patients must have adequate organ and marrow function defined by study-specified laboratory tests.
* For both Women and Men, must use acceptable form of birth control while on study.

Exclusion Criteria:

* Have received any anti-pancreatic cancer therapy.
* Have been diagnosed with another malignancy whose natural history or treatment has the potential to interfere with safety or efficacy assessment of this study.
* Conditions, including alcohol or drug dependence, intercurrent illness, or lack of sufficient peripheral venous access, that would affect the patient's ability to comply with study visits and procedures
* Subjects with active, known or suspected autoimmune disease that may relapse.
* Systemic steroid therapy (> 10mg daily prednisone equivalent) or immunosuppressive therapy within 14 days of first dose of study drug administration.
* Active infection requiring systemic therapy.
* Infection with HIV or hepatitis B or C at screening•
* History of interstitial lung disease, non-infectious pneumonitis or uncontrolled diseases including pulmonary fibrosis, acute lung diseases, etc.
* Uncontrolled intercurrent illness including, but not limited to, uncontrolled infection, pulmonary embolism, uncontrolled hypertension, symptomatic congestive heart failure, unstable angina, cardiac arrhythmia, metastatic cancer, or psychiatric illness/social situations that would limit compliance with study requirements.
* Prior allogeneic stem cell transplantation or organ transplantation
* Any major surgical procedure requiring general anesthesia ≤ 28 days before first dose of study drug.
* Have received a live vaccine ≤ 28 days before first dose of study drug.
* Use of QT prolonging drugs within 2 weeks before the start of SX-682 dosing and for the length of the study.
* ECG demonstrating a QTc interval ≥ 470 msec or patients with congenital long QT syndrome.
* Severe hypersensitivity reaction to any monoclonal antibody.
* Concurrent participation in another therapeutic clinical study
* Pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2023-11-08 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Change in Immune response rate as assessed by density of intratumoral granzyme B+ CD137+ T cells | Baseline and 2 weeks
  The change in density of intratumoral granzyme B+ CD137+ T cells before and after neoadjuvant treatment with tislelizumab and SX-682.
Pathologic Response Rate as assessed by number of patients with a grade 0-2 pathologic response | 4 years
  The number of patients with a grade 0-2 pathologic response as defined by the College of American Pathologists (CAP) tumor regression grading system.

SECONDARY OUTCOMES:
Number of participants experiencing grade 3 or above drug-related toxicities | 4 years
  When calculating the incidence of AEs, each AE (as defined by NCI CTCAE v5.0) will be counted only once for a given subject.
Overall Survival (OS) | 4 years
  OS is defined as the time from the first dose of study treatment to death from any cause. Patients who have not died will be censored at the last date known to be alive. Estimation based on the Kaplan-Meier curve.
Disease Free Survival (DFS) | 4 years
  DFS is defined as the time from the first dose of study treatment until evidence of disease recurrence or death from any cause. For patients who have not progressed, relapsed, or died at the time of analysis, DFS will be censored on the date of last visit where disease progression was evaluable. Estimation based on the Kaplan-Meier curve.

CONTACTS AND LOCATIONS:
Overall Officials: Lei Zheng, MD, Principal Investigator — The University of Texas Health Science Center at San Antonio
Locations (2):
- United States (2):
  - Johns Hopkins SKCCC, Baltimore, Maryland
  - The University of Texas Health Science Center San Antonio, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No